CLINICAL TRIAL: NCT06707259
Title: Clinical Study of Cord Blood-derived IL-10/IL-15 CD19-CAR NK in the Treatment of Refractory/Relapsed B-cell NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024（1369）
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CB IL-10/IL-15-CD19-CAR NK (Experimental): All subjects were intravenously administrated with IL-10/IL-15 CD19-CAR NK
  Interventions: Biological: anti-CD19 IL10/IL15 CAR-NK

INTERVENTIONS:
Biological: anti-CD19 IL10/IL15 CAR-NK — Lentiviral vector-transducted cord blood-derived NK cells to express anti-CD19-IL10/IL-15 CAR

SUMMARY:
To study the safety and effectiveness of cord blood-derived IL-10/IL-15 CD19-CAR NK in patients with B-cell non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
This is an open, single-arm, single-dose, dose-escalation clinical trial designed to evaluate the safety and the preliminary efficacy of CB IL-10/IL-15 CD19-CAR NK cells. 6-24 patients are planned to be enrolled in the dose-escalation trial (2×10^6 cells/kg,4×10^6 cells/kg, 8×10^6 cells/kg). Based on the results in the dose-escalation trial, the recommended dose will be determined. Another 30 patients will be enrolled in the dose-expansion trial. The primary endpoints are DLT and MTD; the second is the overall response rates (CR and PR), survival, and progression-free survival. Patients will be infused on day 0, day 3, and day 6， respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study and sign an informed consent form;
2. Age 18-75 years old, no gender limit;
3. Histologically diagnosed as diffuse large B-cell lymphoma (DLBCL), transforming follicular lymphoma (TFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL) and other inert B-cells NHL conversion type:(1) Refractory or relapsed DLBCL refers to the failure to achieve complete remission after 2-line treatment; disease progression during any treatment, or disease stable time equal to or less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation ； (2) Refractory or relapsed MCL must be resistant to or intolerable to BTK inhibitors; (3) Refractory or relapsed indolent B-cell NHL is the failure or recurrence of third-line treatment; (4) Previous treatment must include CD20 monoclonal antibody treatment (unless the subject is CD20 negative) and anthracyclines;
4. At least one measurable lesion with the longest diameter ≥ 1.5 cm exists;
5. The expected survival period is ≥12 weeks;
6. The puncture section of the tumor tissue was positive for CD19 expression; 7, ECOG score 0-2 points;
7. Sufficient organ function reserve: (1) Alanine aminotransferase, aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value); (2) Creatinine clearance rate (Cockcroft-Gault method) ≥60 mL/min; (3) Serum total bilirubin and alkaline phosphatase ≤1.5× UNL; （4）Glomerular filtration rate>50Ml/min Cardiac ejection fraction (EF) ≥50%; (5) Under natural indoor air environment, basic oxygen saturation>92% .
8. Allow a previous stem cell transplantation.
9. The approved anti-B-cell lymphoma treatments, such as systemic chemotherapy, systemic radiotherapy, and immunotherapy, have been completed for at least 3 weeks before the study medication;
10. Allow patients who have previously received CAR-T cell therapy and have failed or relapsed after 3 months of evaluation;
11. Female subjects of childbearing age must have a negative pregnancy test and agree to take effective contraceptive measures during the trial.
12. Two tests for the new coronavirus were negative.

Exclusion Criteria:

1. Those who have a history of allergies to any of the ingredients in cell products;
2. History of other tumors;
3. Previously presented with II-IV degree (Glucksberg criteria) acute GvHD or extensive chronic GvHD; or are receiving anti-GvHD treatment;
4. Have received gene therapy in the past 3 months;
5. Active infections that require treatment (except for simple urinary tract infections and bacterial pharyngitis), but preventive antibiotics, antiviral and antifungal infection treatments are allowed;
6. Hepatitis B (HBsAg positive, but HBV-DNA <103 is not an exclusion criterion) or hepatitis C virus infection (including virus carriers), syphilis and other subjects with acquired and congenital immunodeficiency diseases, including but not limited to people living with HIV;
7. According to the New York Heart Association's Heart Function Classification Standard, it is classified as Grade III or Grade IV impaired subjects;
8. Those who have received anti-tumor therapy in the early stage but the toxic reaction has not recovered (the CTCAE 5.0 toxic reaction has not recovered to ≤1, except for fatigue, anorexia, and hair loss);
9. Subjects with a history of epilepsy or other central nervous system diseases; 10. Enhanced CT or MRI of the head showed evidence of central nervous system lymphoma;

11. Have any other drugs that target CD19; 12. Women who are breastfeeding and unwilling to stop breastfeeding; 13. Any other situation that the investigator believes may increase the subject's risk or interfere with the test results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, and tolerability, and determine the recommended dosage of cord blood-derived Anti-CD19 IL10/IL15-CAR-NK Cell Therapy for B-cell Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to 2 years
  To determine the anti-tumor effectivity of CB IL-10-CD19-CAR NK
Progression free survival (PFS) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Overall survival (OS) | Up to 2 years
Partial response rate (PR) | Up to 2 years
Overall response rate (ORR) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No